CLINICAL TRIAL: NCT04436419
Title: Immunometabolic Effects of Non-drug Strategies in the Clinical Management of Obesity: Translational Study
Acronym: PPAR-NAPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fauqué (Industry)
Collaborators: Institut Polyclinique de Cannes (IPOCA) (Industry)
Responsible Party: Sponsor-Investigator, Fauqué, Doctor, Institut Polyclinique de Cannes (IPOCA)
Organization: Institut Polyclinique de Cannes (IPOCA) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3573-I
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Obesity, Abdominal; Obesity, Visceral; Female
Keywords: Regulatory T cells; Immunometabolic; Alpha lipoic acid; Physical activity; Non-drug strategy; Obesity
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Motor Activity | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients benefited from a complete hospitalization including dietary monitoring (food intake was controlled in order to provide 30% less of their estimated daily energy expenditure) with a personalized food plan and an adapted physical activity program (5 sessions per week supervised by a graduated health physical activity coach), plus placebo administration (2x per day) apart from meal.
  Interventions: Dietary Supplement: Placebo (full hospitalization: dietary monitoring with an adapted physical activity program)
- ALA (Active Comparator): Patients benefited from a complete hospitalization including dietary monitoring with a personalized food plan and an adapted physical activity program, plus R-ALA enantiomer administration (2x300mg per day) apart from meal.
  Interventions: Dietary Supplement: Alpha lipoic acid (plus full hospitalization)

INTERVENTIONS:
Dietary Supplement: Alpha lipoic acid (plus full hospitalization) — Women are included in an 8-weeks randomized double-blind against placebo supplementation study with ALA (eight per group) according to the following criteria:
  Inclusion criteria: BMI> 30; aged between 18 and 75 years. Non-inclusion criteria: HLA-DRB1*04-03/06 polymorphisms; recent hospitalization (<1 month); food supplement based on antioxidant; medicated in fibrate / telmisartan (modulator of PPARs); patients presenting an acute inflammatory state.
  Exclusion criteria: Pregnant and/or lactating women; not affiliated with social security; not mutual health insurance; person deprived of liberty; participation in clinical research in the last 6 months.
  Patients included in this clinical trial benefited from a complete hospitalization including dietary monitoring with a personalized food plan and an adapted physical activity program. α-LA (2x300mg/day of R-ALA) was administered double-blinded in the form of 2 capsules apart from meals.
  Arms: ALA
Dietary Supplement: Placebo (full hospitalization: dietary monitoring with an adapted physical activity program) — Women are included in an 8-weeks randomized in placebo group. Patients included in this clinical trial benefited from a complete hospitalization including dietary monitoring with a personalized food plan and an adapted physical activity program. Placebo (2x300mg/day) was administered double-blinded in the form of 2 capsules apart from meals.
  Arms: Placebo

SUMMARY:
Forty women aged between 18 and 75 years-old with a BMI> 30kg/m2 are recruited to participate in the evaluation of their medical management. They participate in an 8-week protocol as part of hospital medical treatment for weight loss at the Oxford Polyclinic in Cannes (IPOCA). The effects of 2 independent variables will be studied: (1) an adapted physical activity program and (2) nutritional supplementation with R-α-Lipoic acid (2x300mg/d) versus placebo (double-blind). The volunteers are randomly assigned to the different groups: Placebo with or without exercise groups and ALA with or without exercise groups. At the start of the protocol (T0), at 4 weeks (T4) and at 8 weeks (T8), various measurements are carried out (physical capacities, nutritional status, body composition, distribution of adipose mass by CT-scan). A venous sample taken for all participants is done at T0, T4 and T8 to investigate the immune profile of circulating T lymphocytes.

This project is part of a translational research project to assess current care and to investigate the immunometabolic effects of a non-drug medical care of obesity (adapted physical activities, nutritional supplementation with α-lipoic acid, quality of food intake).

DETAILED DESCRIPTION:
Obesity-related inflammation is central to the development of type 2 diabetes and potentiated by advancing age, inactive behavior and sedentary lifestyle. Metabolism and immunity are entangled in their respective effects: the pathways of inflammation are involved in metabolism and the metabolic state plays a predominant role in immune function. Physical activity and calorie restriction are first-line, non-drug strategies recommended in reducing obesity and insulin resistance and then prevent type 2 diabetes. However, the impact of their combined effects on circulating immune cells or those residing in adipose tissue and skeletal muscle, remains insufficiently understood to allow a nutritional prescription (i.e., quality of nutritional intake and efficient doses of physical activity) favorable to preventive medical care, individualized, and effective. If the risk associated with an increase in visceral fat mass is linked to a change in the pro/anti-inflammatory status, it is essential to reduce this risk by acting on its cause, regardless of the weight loss. In a context of low-grade inflammation, these effects could lead to an anti-inflammatory profile of T cells, specifically regulatory T cells (Treg) whose metabolism is extremely "flexible" at the periphery and into visceral adipose tissue (directly involved in inflammation of obesity).

ALA (Alpha-Lipoic Acid) is known to play a pivotal role in cellular redox status and energy metabolism by modulating inflammatory and metabolic signaling pathways such as those of NF-kB, JNK, PI3K/Akt, p38 MAPK, AMPK or PPARβ/δ. As ALA is a possible metabolic modulator, it would affect the metabolism of T cells. And therefore ALA could be a complementary measure to non-drug strategies by potentiating the correction of the inflammatory state linked to obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 30; aged between 18 and 75 years

Exclusion Criteria:

* Pregnant and/or lactating women; not affiliated with social security; not mutual health insurance; person deprived of liberty; participation in clinical research in the last 6 months

Non-inclusion criteria:

* HLA-DRB1*04-03/06 polymorphisms; recent hospitalization (<1 month); food supplement based on antioxidant; medicated in fibrate/telmisartan (modulator of PPARs)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Variation in the prevalence of regulatory T cells from Peripheral Blood Mononuclear Cells (PBMCs) drawn from whole blood at the beginning (T0), mid-course (T4) and the end of the course (T8). | Through study completion, an average of 2 months
  Cells were gently washed twice and resuspended in PBS. Stained cell preparations were analyzed using a BD FACS Canto II flow cytometer. The staining and gating strategy were used for traited human PBMCs by utilizing CD3+, CD4+, CD25+ and FoxP3+ antibodies. We have discriminated CD3+CD4+ versus CD3+CD4-. Finally, at this stage CD25+FoxP3+ (Regulatory T cells) cells were gated as part of the CD3+CD4+ population.
60% increasing in PPARβ/δ expression, estimated from the level of expression of its main target gene CPT1a, in human PBMC between the beginning (T0) and end of the course (T8). | Through study completion, an average of 2 months
  Total mRNA was extracted with Trizol reagent and the relative amount of CPT1a mRNA was calculated using the comparative ΔΔCT method after quantitative RT-PCR analysis.
Improvement of Redox status by measuring GSH/GSSH ratio in human whole blood between the beginning (T0) and end of the course (T8). | Through study completion, an average of 3 months
  The GSH/GSSG Assay is designed to accurately measure total, reduced and oxidized glutathione in biological samples using an enzymatic method that utilizes Ellman's Reagent (DTNB) and glutathione reductase (GR).

SECONDARY OUTCOMES:
Reduction of the area from visceral adipose tissue measured by computed-tomography scan between the beginning (T0) and end of the course (T8). | Through study completion, an average of 1 months
  A computed-tomography scan (CT-scan) which allowed to discriminate the area of subcutaneous adipose tissue from visceral fatty area (VFA) was calculated from x-ray performed at the third lumbar level. Visceral abdominal adipose tissue was estimated by subtracting total abdominal and subcutaneous adipose tissues areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinic of Oxford (IPOCA), Cannes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gleeson M, Bishop NC, Stensel DJ, Lindley MR, Mastana SS, Nimmo MA. The anti-inflammatory effects of exercise: mechanisms and implications for the prevention and treatment of disease. Nat Rev Immunol. 2011 Aug 5;11(9):607-15. doi: 10.1038/nri3041. PMID 21818123
- [Background] Mothe-Satney I, Murdaca J, Sibille B, Rousseau AS, Squillace R, Le Menn G, Rekima A, Larbret F, Pele J, Verhasselt V, Grimaldi PA, Neels JG. A role for Peroxisome Proliferator-Activated Receptor Beta in T cell development. Sci Rep. 2016 Sep 29;6:34317. doi: 10.1038/srep34317. PMID 27680392
- [Background] Rousseau AS, Sibille B, Murdaca J, Mothe-Satney I, Grimaldi PA, Neels JG. alpha-Lipoic acid up-regulates expression of peroxisome proliferator-activated receptor beta in skeletal muscle: involvement of the JNK signaling pathway. FASEB J. 2016 Mar;30(3):1287-99. doi: 10.1096/fj.15-280453. Epub 2015 Dec 9. PMID 26655383
- [Background] Le Garf S, Murdaca J, Mothe-Satney I, Sibille B, Le Menn G, Chinetti G, Neels JG, Rousseau AS. Complementary Immunometabolic Effects of Exercise and PPARbeta/delta Agonist in the Context of Diet-Induced Weight Loss in Obese Female Mice. Int J Mol Sci. 2019 Oct 19;20(20):5182. doi: 10.3390/ijms20205182. PMID 31635041
- [Background] Namazi N, Larijani B, Azadbakht L. Alpha-lipoic acid supplement in obesity treatment: A systematic review and meta-analysis of clinical trials. Clin Nutr. 2018 Apr;37(2):419-428. doi: 10.1016/j.clnu.2017.06.002. Epub 2017 Jun 8. PMID 28629898
- [Background] Cui J, Huang D, Zheng Y. Ameliorative effects of alpha-lipoic acid on high-fat diet-induced oxidative stress and glucose uptake impairment of T cells. Free Radic Res. 2016 Oct;50(10):1106-1115. doi: 10.1080/10715762.2016.1210140. Epub 2016 Aug 4. PMID 27383289
- [Background] Berod L, Friedrich C, Nandan A, Freitag J, Hagemann S, Harmrolfs K, Sandouk A, Hesse C, Castro CN, Bahre H, Tschirner SK, Gorinski N, Gohmert M, Mayer CT, Huehn J, Ponimaskin E, Abraham WR, Muller R, Lochner M, Sparwasser T. De novo fatty acid synthesis controls the fate between regulatory T and T helper 17 cells. Nat Med. 2014 Nov;20(11):1327-33. doi: 10.1038/nm.3704. Epub 2014 Oct 5. PMID 25282359
- [Background] Kempkes RWM, Joosten I, Koenen HJPM, He X. Metabolic Pathways Involved in Regulatory T Cell Functionality. Front Immunol. 2019 Dec 3;10:2839. doi: 10.3389/fimmu.2019.02839. eCollection 2019. PMID 31849995
- [Background] Newton R, Priyadharshini B, Turka LA. Immunometabolism of regulatory T cells. Nat Immunol. 2016 May 19;17(6):618-25. doi: 10.1038/ni.3466. PMID 27196520
- [Background] Zou J, Lai B, Zheng M, Chen Q, Jiang S, Song A, Huang Z, Shi P, Tu X, Wang D, Lu L, Lin Z, Gao X. CD4+ T cells memorize obesity and promote weight regain. Cell Mol Immunol. 2018 Jun;15(6):630-639. doi: 10.1038/cmi.2017.36. Epub 2017 Jun 19. PMID 28626237